CLINICAL TRIAL: NCT07340593
Title: A Community-based Collaborative Study for Eradication of Helicobacter Pylori and Associated Gastric Cancer in Luangprabang and Champasak Province, in Lao PDR 2025.
Brief Title: Helicobacter Pylori Infection and Gastric Diseases in Lao PDR: First Community-Wide Population-Based Study
Status: Completed | Type: Observational
Sponsor: Zero Helicobacter IGAN Network (Other)
Collaborators: Oita University (Other); Setthathirath Hospital (Other); Mahosot Hospital, Laos (Unknown); Lao National Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 1015/REC
Record Dates: First submitted 2025-12-19; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer Screening; Prevention and Control; Helicobacter Eradication; Helicobacter Infections
Keywords: gastric cancer; helicobacter pylori; Laos; H pylori eradication; cancer prevention
MeSH Terms: conditions — Helicobacter Infections; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gastric biopsy samples for molecular analysis of antimicrobial resistance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Residents of Luang Prabang Province: Residents aged ≥18 years in Luang Prabang Province who underwent stool antigen testing for H. pylori.
  Participants ≥40 years who tested positive additionally underwent upper endoscopy.
  All positive individuals received triple therapy and were followed for eradication.
- Residents of Champasak Province: Residents aged ≥18 years in Champasak Province who underwent stool antigen testing for H. pylori.
  Participants ≥40 years who tested positive additionally underwent upper endoscopy.
  All positive individuals received triple therapy and were followed for eradication.

SUMMARY:
This study aims to determine the regional prevalence of Helicobacter pylori infection, bacterial strain differences, and the prevalence of gastric cancer in two provinces of Laos, a multi-ethnic country where these factors may vary by region and ethnicity. The study also evaluates whether H. pylori eradication therapy contributes to disease prevention. Residents aged 18 years or older in Luang Prabang Province and Champasak Province underwent stool antigen testing, and H. pylori-positive individuals received eradication therapy. High-risk participants aged ≥40 years underwent upper gastrointestinal endoscopy for early detection of gastric cancer.

DETAILED DESCRIPTION:
This population-based study was conducted in Laos to investigate geographic variation in Helicobacter pylori infection, bacterial strains, and the prevalence of precancerous and cancerous gastric lesions. Laos is a multi-ethnic nation, and differences in H. pylori prevalence and strain distribution are expected across ethnic groups and regions. The goal of this study is to assess the current burden of infection and evaluate the effectiveness of eradication therapy as a preventive strategy for gastric cancer.

Eligible participants were residents aged ≥18 years living in Luang Prabang Province (North) and Champasak Province (South). The study received approval from the Ethics Committee of the Ministry of Health of Laos. All participants received an explanation of the risks and benefits of screening and provided written informed consent.

The study procedures were conducted as follows:

1. Stool H. pylori antigen rapid test was performed for all enrolled participants.
2. Participants aged ≥40 years who tested positive were considered a high-risk group and underwent upper gastrointestinal endoscopy for early detection of precancerous gastric lesions and gastric cancer.
3. All H. pylori-positive participants received 14-day triple therapy consisting of lansoprazole, amoxicillin, and clarithromycin.
4. Eradication was assessed using a follow-up stool antigen test at 8 months after treatment in Luang Prabang Province and 6 months after treatment in Champasak Province.

Screening in Luang Prabang Province was conducted between December 2023 and October 2024, and screening in Champasak Province between October 2024 and June 2024.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Resident of Luangprabang or Champasak Province
* Able to provide written informed consent

Exclusion Criteria:

* Severe comorbidities contraindicating screening or treatment
* Allergy to medications used in triple therapy
* Pregnant or breastfeeding women (if applicable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study Locations
  1. Luangprabang Province, Lao PDR
  2. Champasak Province, Lao PDR
Sampling Method: Non-Probability Sample
Enrollment: 1251 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-06-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of H. pylori infection • Method: Stool antigen test • Time Frame: Baseline | Baseline
  The proportion of participants who test positive for H. pylori infection using a stool antigen rapid test at baseline.
  All enrolled residents aged ≥18 years in Luang Prabang Province and Champasak Province undergo stool antigen testing. H. pylori positivity is defined according to the manufacturer's validated cutoff value.
  This measure provides a population-based estimate of the current H. pylori infection prevalence in two geographically distinct regions of Laos.

SECONDARY OUTCOMES:
H. pylori eradication rate after triple therapy, | 6-8 months after treatment completion,
  The percentage of H. pylori-positive participants who achieve eradication following 14-day triple therapy, confirmed by stool antigen testing.

OTHER OUTCOMES:
Prevalence of gastric cancer | Baseline endoscopy
  Number of gastric cancer detected during screening endoscopy among high-risk participants (≥40 years, H. pylori positive).

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Vientiane, Capital, Laos

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Due to ethical and regulatory considerations in Laos, and because the dataset includes sensitive health information collected from community residents, de-identified participant-level data will not be made publicly available.